CLINICAL TRIAL: NCT00981513
Title: Direct and Indirect Benefits of Influenza Vaccination in Schools and Households
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Dr Benjamin J. Cowling, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BJC004.6
Record Dates: First submitted 2009-09-20; First posted 2009-09-22 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-08

CONDITIONS: Influenza Virus Infection; Influenza-like Illness; Acute Respiratory Infection
MeSH Terms: interventions — FluMist; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Influenza vaccination (Active Comparator): Live attenuated influenza vaccine (seasonal and pandemic strains) by nasal spray
  Interventions: Biological: Trivalent live attenuated seasonal influenza vaccine; Biological: Monovalent live attenuated pandemic influenza vaccine
- Saline placebo (Placebo Comparator): Saline nasal spray
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: Trivalent live attenuated seasonal influenza vaccine — One dose
  Other Names: FluMist, MedImmune Vaccines, Inc.
  Arms: Influenza vaccination
Biological: Monovalent live attenuated pandemic influenza vaccine — One dose
  Other Names: FluMist Novel H1N1, MedImmune Vaccines, Inc.
  Arms: Influenza vaccination
Biological: Saline — One dose
  Other Names: Saline nasal spray
  Arms: Saline placebo

SUMMARY:
The purpose of this study is to determine the degree of indirect benefits to family members and classmates resulting from administration of influenza vaccine to children.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged between 7 and 11 and their family members.

Exclusion Criteria:

* Children with history of hypersensitivity to eggs, egg proteins, gentamicin, gelatin, or arginine or with life-threatening reactions to previous influenza vaccinations.
* Children receiving aspirin therapy or aspirin-containing therapy.
* Children with asthma or active wheezing.
* Children or family members with underlying immunocompromised condition or receiving immunosuppressive agents.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6300 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Clinical influenza by self-reported symptoms, specifically defined as at least two of fever ≥37.8ºC, cough, headache, sore throat, aches or pains in muscles or joints | One year
Influenza virus infection confirmed by RT-PCR | One year

SECONDARY OUTCOMES:
Influenza virus infection during the follow-up period assessed by four-fold or greater rise in paired serology. | One year
Adverse events following vaccination | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Cowling, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Pokfulam, Hong Kong